CLINICAL TRIAL: NCT05301777
Title: Computed Tomography Anatomy of the Paranasal Sinuses and Anatomical Variants of Clinical Relevants in Egyptian Adults .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Emad Eldin Moghazy, Assuit university radiology department, Assiut University
Other Study IDs: CT paranasal sinuses
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Computed tomography — Computed tomography

SUMMARY:
The aim of this study is to show the anatomy of the paranasal sinuses as delineated by the computed tomography among egyptian adults and to describe the variants which not only predispose to chronic sinusitis but may lead to complications in endoscopic sinonasal surgery.

DETAILED DESCRIPTION:
The paranasal sinuses are group of air filled spaces surrounding the nasal cavity; which start developing from the primitive choana at 25-28 weeks of gestation.1 Three projections arise from the lateral wall of the nose and serve as the beginning of the development of the paranasal sinuses. The anterior projection forms the Aggernasi, the inferior or maxiloturbinate projection forms the inferior turbinates and maxillary sinus, while the superior or ethmoidoturbinate projection forms the ethmoidal air cells and their corresponding drainage channels. The sinuses are named from the facial bones in which they are located. The maxillary and ethmoid sinuses are aerated at birth, while the sphenoid sinuses and frontal sinuses are pneumatized at about the 2nd and 6th year of life respectively.1 The sinuses reach the adult size at adolescent age.1 Radiologic evaluation of the paranasal sinuses is essential in delineating the location and extent of sinonasal diseases and in planning surgical intervention. Plain radiography, computed tomography and magnetic resonance imaging are applied in evaluating the sinuses.

Standard paranasal sinus radiograph can readily demonstrate the maxillary or frontal sinus diseases but incompletely delineates ethmoid sinus due to overlapping of structures.2 The role of Magnetic resonance imaging is limited but may provide information on paranasal sinuses fungal infection and differentiating thickened mucosa from fluid retention.

Computed tomography is considered the method of choice in delineating completely the normal anatomy and anatomical variants of the paranasal sinuses and it is extremely useful in the pre-operative planning and in post operative follow-up in cases of endonasal interventions.

The development of the paranasal sinuses especially the ethmoid labyrinth is associated with anatomical variations.3 Some of which are common while others are rare. Recognition of these variants is important to both the rhinologist and radiologist. Proximity of these occasional cells to the main drainage pathway of the paranasal sinuses may reduce the mucociliary clearance, thus predisposing to inflammatory processes and causing endonasal endoscopic surgery complications.

ELIGIBILITY:
Inclusion Criteria:

* all cases of computed tomography scan of the paranasal sinuses obtained in the Radiology department of our health institution

Exclusion Criteria:

* Patients with facial trauma, positive paranasal sinus pathology, head and neck tumours

and previous surgery were excluded.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
show the anatomy of the paranasal sinuses as delineated by the computedtomography and | Baseline
  show the anatomy of the paranasal sinuses as delineated by the computedtomography and to describe the variants which not only predispose to chronic sinusitis but may lead to complications in endoscopic sinonasal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Hashem, Principal Investigator — Assiut University; Hazem Abozaid, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
CT anatomy of paranasal sinuses in egyptian adults
Supporting Information: Study Protocol
Time Frame: In 2 years
Access Criteria: Para nasal sinuses
URL: http://www.sciencedirect.com/science/article/pii/S2090074016300688